CLINICAL TRIAL: NCT04466982
Title: Objective Assessment of Olfactory Dysfunction and Impact on Quality of Life in SARS CoV-2 (COVID-19)Infection Using the UPSIT, eQOD and SNOT-22 Questionnaires: A Prospective Observational Cohort Study
Brief Title: Assessment of Olfactory Dysfunction in SARS CoV-2 (COVID-19) Infection
Acronym: ODYSSI
Status: Completed | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other); Royal Cornwall Hospitals Trust (Other)
Responsible Party: Principal Investigator, Ekpemi Irune, Consultant in Otolaryngology, Head & Neck Surgery, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: REC Ref: 20/SC/0231
Record Dates: First submitted 2020-07-09; First posted 2020-07-10 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Olfactory Disorder; COVID19; SARS-CoV-2; Anosmia; Microsomia; Smell Disorder; Quality of Life
MeSH Terms: conditions — COVID-19; Anosmia; Fetal Growth Retardation; Olfaction Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is designed to investigate the acuity of olfactory dysfunction in COVID-19 positive patients in the United Kingdom. In particular defining severity with objective testing and determining if this has any predictive value on the outcome of the SARS CoV-2 infection. In addition, this study will strive to determine duration / natural history of olfactory dysfunction in these patients in respect to a positive SARS CoV-2 diagnosis. It should also demonstrate the impact of olfactory dysfunction on patient Quality of Life (QOL).

DETAILED DESCRIPTION:
The main objective of this study is to evaluate olfactory acuity by means of a multidimensional assessment protocol to objectively demonstrate the severity of olfactory dysfunction in patients diagnosed with SARS CoV-2. The University of Pennsylvania Smell Identification Test (UPSIT) will be used to assess olfactory function in newly diagnosed patients and also existing patients longitudinally over a 12-month period. This is to document onset (where possible) and rate of progress of olfactory dysfunction.

In relevant cases, the investigators will correlate their findings with severity of the Acute Respiratory Distress Syndrome (ARDS) arising as a result of the infection - characterised as mild, moderate and severe according to the Berlin classification. The investigators will therefore determine if the degree of olfactory dysfunction correlates in any manner to the severity of ARDS developed in a positive SARS CoV-2 patient and if it offers any prognosticative applications.

The investigators will also examine the impact of the symptom of olfactory dysfunction on patient Quality of Life using two validated tools known as the Questionnaire of Olfactory Disorders for English speakers (eQOD) and the SNOT-22 questionnaire.

Furthermore, outcomes will be explored and stratified in terms of age, gender and ethnicity

ELIGIBILITY:
Inclusion Criteria:

* Patients who are presenting to hospital with symptoms of SARS CoV-2 infection.
* Patients who go on to develop a positive SARS CoV-2 test.
* Patients who can give a valid written informed consent.
* Patients who are motivated to participate in the study.
* Adult patients aged 18 years - 85 years.

Exclusion Criteria:

* Patients who cannot give a valid written informed consent.
* Patients who are not willing or not motivated to participate in the study.
* Patients with negative SARS CoV-2 tests.
* Patients with nasal pathologies like severe deviated nasal septum, nasal masses, head trauma or previously known chronic rhinosinusitis with polyps or on medication for more than 6 months/year for at least one year for chronic rhinosinusitis.
* Patients with any diagnosed neurological disease known to affect olfactory function will be excluded from the study.
* Patients unable to read in the English language.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study group will comprise patients diagnosed with the SARS Cov-2 infection at the local site.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
UPSIT scores | At time of diagnosis (+1 week ) post COVID 19 diagnosis or at time of recruitment into study
  I. Primary endpoint is olfactory function assessed using the UPSIT and classified as Anosmia; Mild, moderate, and severe microsomia. assessed at the time COVID-19 diagnosis (+1 week) or at the time of registration for in hospital patients

SECONDARY OUTCOMES:
UPSIT scores | at day 0, 1 month, 3 month, 6 month, 9 month and 12 month
  I. The changes in olfaction in patients with SARS CoV-2 infection over an initial 12 month period (at day 0, 1 month, 3 month, 6 month, 9 month and 12 month) using the UPSIT.
eQOD scores | at day 0, 1 month, 3 month, 6 month, 9 month and 12 month
  Quality of Life using the validated Questionnaire of Olfactory Disorders for English speakers (eQOD)
SNOT 22 scores | at day 0, 1 month, 3 month, 6 month, 9 month and 12 month
  Quality of Life using the validated SinoNasal Outcome Tool-22 (SNOT-22)

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Addenbrookes Hospital, Cambridge
  - Charing Cross Hospital, London
  - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: No